CLINICAL TRIAL: NCT07043738
Title: Imaging- vs. Scalp-Targeted Accelerated TMS for Depression: The Number Needed to Scan Trial
Acronym: NNS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joseph J. Taylor, MD, PhD, Assistant Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P001570
Record Dates: First submitted 2025-06-26; First posted 2025-06-29 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Accelerated Transcranial Magnetic Stimulation; Depression; Major Depressive Disorder; Treatment resistant depression; TMS; Transcranial Magnetic Stimulation; Neuromodulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel-group double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study participants will get two treatment sites marked: 1) Their individualized target based on resting state functional connectivity data, and 2) Beam F3 target based on head measurements. One group will be treated at target #1, and the other group will be treated at target #2. The research assistant (RA) marking treatment sites is the only individual unblinded in this study. The unblinded RA will have no other interactions with participants after the treatment preparation visit. RAs delivering treatment with stimulate participants at a coordinate, given to them by the unblinded RA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Connectivity-based targeting (Other): Participants in this group will receive aiTBS with neuronavigation to a treatment target identified with individualized resting state functional connectivity.
  Participants who receive connectivity-based targeting and who do not meet response criteria (<50% MADRS improvement) at the post-treatment month 1 visit will be offered the opportunity to opt in and receive another course of aTMS at their scalp-based target.
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Scalp-based targeting (Other): Participants in this group will receive aiTBS with neuronavigation to a treatment target identified with scalp based measurements (i.e., Beam F3).
  Participants who receive scalp-based targeting and who do not meet response criteria (<50% MADRS improvement) at the post-treatment month 1 visit will be offered the opportunity to opt in and receive another course of aTMS at their connectivity-based target.
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a focal, non-invasive form of brain stimulation that has FDA clearance for depression. In this study, a form of TMS called accelerated intermittent theta burst stimulation (aiTBS) will be administered under the supervision of a physician with TMS expertise.
  Other Names: TMS; Accelerated intermittent theta burst stimulation; aiTBS

SUMMARY:
Transcranial magnetic stimulation(TMS) is a non-invasive form of brain stimulation that is cleared by the United States Food and Drug Administration (FDA) for depression. Conventional TMS involves daily weekday treatments for 6-8 weeks. These treatments are targeted using each person's scalp measurements. With conventional TMS, approximately 50-55% of people show a 50% or more improvement in depressive symptoms (in other words, they "respond" to treatment).

Studies are trying to make TMS work better and faster. A new form of TMS called accelerated TMS (aTMS) involves mutliple treatments a day. One specific aTMS protocol involves 10 treatments per day for 5 days. These treatments are targeted using each person's brain scan (magentic resonance imaging, MRI). With this specific aTMS protocol, approximately 70-90% of people show a 50% or more imporvement in depressive symptoms. While these results are exciting, scientists are not sure why this specific aTMS protocol works better than conventional TMS. It could be the dose and schedule of treatment, or it could be the MRI-based targeting. Answering this question is important because MRI-based targeting is expensive and difficult to do in many settings.

This study aims to determine if MRI-based targeting is better than scalp-based targeting for aTMS for depression. In this study, everyone who enrolls and meets criteria will be randomly assigned to MRI- versus scalp-based aTMS targeting.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) remains a leading cause of global disease burden and disability. In addition to increasing the risk of death by suicide, MDD also shows a graded positive association with all-cause mortality. Antidepressants are the most frequently prescribed medication class in psychiatry and, once started, are often continued for many year. However, antidepressants have a small-to-moderate effect size that might be inflated by publication bias. Most people with MDD do not achieve remission with their first antidepressant, and the probability of getting well and staying well diminishes with each sequential trial. By the fourth trial, remission rates approach single digits. Depression that does not improve with one or more antidepressant classes is often considered "difficult-to-treat" or "treatment-resistant" depression (TRD). Taken together, these data highlight the need for better and faster treatments for TRD.

TMS for TRD is safe, well-tolerated, and often covered by insurance. Unlike esketamine and ECT, TMS does not require supervised transportation after treatment. However, TMS is: 1) time intensive, requiring daily weekday treatments for 6-8 weeks; 2) imprecisely targeted based on scalp measurements, which means that each person is stimulated at a slightly different site; and 3) ineffective approximately half the time, with response and remission rates around 50% and 33%, respectively. A new form of accelerated TMS (aTMS) by Cole et. al was designed to address these limitations. In the open-label trial (n=21), the Cole et a. protocol significantly reduced Montgomery-Åsberg Depression Rating Scale (MADRS) in a single day and resulted in a 79.5% reduction one month after treatment. Remission rates were 86% and 57% one week and one month after open-label aTMS, respectively. From this perspective, this specific aTMS protocol works better and faster than conventional TMS and even rivals ECT. The only double-blind randomized controlled trial of this Cole et al. protocol was discontinued after an interim analysis (n=29) revealed a large effect size (Cohen's d>0.8) for active vs. sham (52.5% vs. 11.1% MADRS reduction, respectively). In this trial, remission rates were 57% and 46% one week and month after active aTMS, respectively. There are also emerging data on retreatment and durability. In a recent open-label extension study (n=27), 91% of people who achieved remission with an index course of this specific aTMS protocol (n=22) also achieved remission with aTMS retreatment 6 months later.

In July 2023, investigators launched the "AINT Trial" (NCT05680727). Our goal was to calculate an effect size to power a confirmatory trial. Investigators matched Cole et al. on schedule, dose, intensity, and precision. Investigators also matched Cole et al. inclusion/exclusion criteria (based on published trials and feedback from Stanford colleagues) and its primary outcome measure (i.e., MADRS reduction (% change) one month after aTMS). The goal was to isolate the variable of targeting. Based on our results (in preparation), a sample size of 40 per group will provide ~95% power to detect a between-group difference. Therefore, this study will be a fully powered, double-blind, confirmatory efficacy trial (n=80) for imaging- vs. scalp-targeted aTMS for TRD.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-80
* English proficiency sufficient for informed consent, questionnaires/tasks, and treatment
* Primary diagnosis of major depressive disorder per DSM-V criteria (Quick Structured Clinical Interview for DSM-5)

  * >20 on Beck Depression Inventory (BDI)
  * >20 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
  * Moderate to severe level of treatment resistance (Maudsley Staging Method)
* Stable antidepressant medication regimen, or remain medication free, for 4 weeks prior to treatment and to remain on this regimen throughout the study until the 1-month post-treatment visit.
* Primary clinician (e.g. psychiatrist, therapist, psychologist, APRN, PA, etc.) responsible for psychiatric care before, during, and after the trial
* Agreement to lifestyle considerations

  * Abstain from becoming pregnant from screening to one-month after treatment (the MRI visit)
  * Continue usual intake patterns of caffeine- or xanthine-containing products (e.g. coffee, tea, soft drinks, chocolate) throughout treatment
  * Abstain from alcohol, tobacco, and recreational drugs for at least 24 hours before the start of each MRI and TMS session

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline to one month post treatment
  Depression severity rating scale (0-60, higher numbers indicate higher depressive symptom severity). The MADRS is a clinician rated scale consisting of 10 items, with each item scored on a 7 point scale.
  For the primary outcome, investigators will assess MADRS as a continuous variable (i.e., MADRS change from baseline to one month after treatment) using a mixed-effects model for repeated measures (MMRM). The model will include group assignment, baseline MADRS score, assessment time point, and time point by treatment interaction as explanatory variables.
  Hypothesis: There will be a significant group x time interaction on MADRS score from baseline, immediately post-treatment (Day 5), one-week post-treatment, and one-month post-treatment.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline to one month post treatment
  Depression severity rating scale (0-60, higher numbers indicate higher depressive symptom severity). The MADRS is a clinician rated scale consisting of 10 items, with each item scored on a 7 point scale. For the secondary outcomes, investigators will assess MADRS as a categorical variable (i.e., MADRS response defined as ≥ 50% improvement one month after treatment) using a generalized estimating equations approach (GEE).
  Hypothesis: One month after treatment, there will be a significantly larger response rate (≥ 50% MADRS improvement) in the imaging- vs. scalp-targeted group using a z-test for proportions. This response rate will be used to calculate an absolute risk reduction and a "number needed to scan" (NNS) with confidence intervals.
Relationship between treatment target location and response in scalp-targeted aTMS for MDD | Before treatment to 1 month post treatment
  The correlation between clinical improvement (i.e., BDI-II) and the distance between the actual (stimulated) scalp-based target and the (predicted but not stimulated) imaging-based target. The BDI-II is a depression severity rating scales (0-63, higher numbers indicate higher severity).
  Mediation analyses that includes the mediator variable (i.e., distance) in the multivariable model for the outcome (i.e., MADRS improvement). Investigators will implement a form (i.e., counterfactual-based) causal mediation analysis that estimates the controlled direct and indirect effects and the bias-corrected bootstrap confidence intervals while controlling for confounders such as age, sex, and other related variables (e.g., baseline antidepressant use, etc.).
  Hypothesis: In the scalp-targeted aTMS group, clinical improvement will negatively correlate with the distance between the actual (stimulated) scalp-based target and the (predicted but not stimulated) imaging-based target.

OTHER OUTCOMES:
Beck Depression Inventory (BDI) | Before treatment, daily throughout treatment, 1 week post treatment, and 1-12 months post treatment
  Depression severity rating scales (0-63, higher numbers indicate higher severity)
Beck Anxiety Inventory (BAI) | Before treatment, daily throughout treatment, 1 week post treatment, and 1-12 months post treatment
  Anxiety severity rating scale (0-63, higher numbers indicate higher severity)
Clinically Useful Depression Outcome Scale - Daily Adaptation (CUDOS-D) | Before treatment, daily throughout treatment, 1 week post treatment, and 1 month post treatment
  Depression severity rating scales (0-64, higher numbers indicate higher severity)
Clinically Useful Anxiety Outcome Scale - Daily Adaptation (CUXOS-D) | Before treatment, daily throughout treatment, 1 week post treatment, and 1 month post treatment
  Anxiety severity rating scale (0-80, higher numbers indicate higher severity)
Patient Global Impression of Change (PGIC) | Before treatment to 1 month post treatment
  A single question assessing a patient's perception of their health or condition (scores range from 1-7, one being the participant believes they are not at all ill, seven being an extremely ill individual) and rate their overall change in condition (scores range from 1-7, one being very much improved and seven being very much worse).
Visual Analog Scale (Mood) | Baseline (before treatment), throughout treatment, and 1 month post treatment
  A single question asking participants to rate their current mood on a scale of 1-100 (higher scores indicate positive mood)
DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure-Adult (DSM-5-XC) | Baseline (before treatment) to 1 month post treatment
  Transdiagnostic rating scale (each question rated 0-4) Minimum score: 0 Maximum score: 92 Higher score indicates worse outcome or worse overall psychiatric burden
Adult Attention Deficit/Hyperactivity Disorder Self-Report Scale (AARS) | Baseline (before treatment) to 1 month post treatment
  ADHD rating scale (each question rated 1-5, higher scores indicate symptoms highly consistent with ADHD)
Illness Intrusiveness Rating Scale (IIRS) | Baseline (before treatment) to 1 month post treatment
  13 item scale measuring how illness affects function. Scored 13-91, higher score indicates higher illness intrusiveness severity
McLean Screening Instrument for Borderline Personality Disorder (MS-BPD) | Baseline (before treatment) to 1 month post treatment
  10-item questionnaire used to screen for BPD (scores range from 0 to 10; higher scores are associated with higher levels of/more severe BPD symptoms).
Perceived Stress Scale (PSS) | Baseline (before treatment) to 1 month post treatment
  Stress assessment scored 0-40, higher scores indicate higher stress
Self-Compassion Scale (SCS) | Baseline (before treatment) to 1 month post treatment
  Scale for assessing self compassion (scores range from 1-5, with higher scores indicating greater well-being).
Social Readjustment Rating Scale (SRRS) | Baseline (before treatment) to 1 month post treatment
  A tool used to assess the potential stress associated with different life events (scores range from 0 to 430, with higher scores indicating higher levels of stress).
Spiritual Transcendence Scale (STS) | Baseline (before treatment) to 1 month post treatment
  24 items with responses ranging from 1 to 5; a higher score would indicate a higher level of spiritual transcendence.
Young Mania Rating Scale (YMRS) | Before treatment, throughout treatment, to 1 month post treatment
  11 item scale evaluating mania. Scored 0-60. Higher score indicates worse outcome/higher mania
World Health Organization Quality of Life (WHOQOL-BREF) | Baseline (before treatment) to 1 month post treatment.
  26-item questionnaire assessing an individual's perception of their quality of life (scores range from 0 to 100, where higher scores represent a better quality of life).
World Health Organization Disability Assessment Schedule II (WHODAS 2.0) | Baseline (before treatment) to 1 month post treatment
  36-item functional assessment (each question rated 1-5) Minimum: 36 Maximum: 180 Can also be scored by percentiles Higher score indicates more disability
Death-Suicide Implicit Association Task | Baseline (before treatment) to 1 month post treatment
  Computer task measuring reaction time
Emotion Conflict Resolution (ECR) | Baseline (before treatment) to 1 month post treatment
  Computer task measuring accuracy and reaction time to emotional faces
Multisource Interference Task (MSIT) | Baseline (before treatment) to 1 month post treatment
  Computer task measuring accuracy and reaction time
Penn Emotion Recognition Task (ER-40) | Baseline (before treatment) to 1 month post treatment
  Computer task measuring accuracy and reaction time to emotional faces
Tinnitus Handicap Inventory (THI) | Baseline (before treatment) to 1 month post treatment
  25-item self-report questionnaire used to assess the impact of tinnitus on a person's daily life (scores range from 0 to 100; higher scores indicate a greater tinnitus handicap impact)
Anxiety Sensitivity Index (ASI) | Baseline (before treatment) to 1 month post treatment
  16-item self-report questionnaire used to assess the degree to which individuals fear the physical sensations associated with anxiety (scores range from 0 to 64; higher scores indicate greater anxiety sensitivity).
Adult Temperament Questionnaire (ATQ) | Baseline (before treatment) to 1 month post treatment
  77-item self-administered questionnaire that measures the constructs of effortful control, negative affect, extraversion/surgency, and orienting sensitivity (higher scores indicate presence of listed temperament characteristics).

IPD SHARING:
Plan to Share IPD: Undecided